CLINICAL TRIAL: NCT05773131
Title: Remote Cross-Platform VR Collaboration System for Mechanically Ventilated ICU Patients to Improve Mental Health Outcomes
Brief Title: VR Collaboration System to Improve Mental Health Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-3575-1
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-06

CONDITIONS: Mental Health Issue
Keywords: ICU; mechanically ventilated patients; virtual reality; mental health; social connection
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR collaborative visualization group (Experimental): In this intervention system, the stimulation materials, communication interface, collaboration tasks, and immersive 360-degree scenario will be played inside a commercially available head-mounted display on the patient side, as well as these materials will be played in the smartphone on the family members' side.
  Interventions: Device: VR collaborative visualization system
- Standard ICU Care (No Intervention): Patients will be treated with standard ICU care and not receive VR stimulation.

INTERVENTIONS:
Device: VR collaborative visualization system — Patients wear virtual reality head-mounted displays while family members using smart phones to interact in a same virtual space.
  Arms: VR collaborative visualization group

SUMMARY:
Collaboration between family members and mechanically ventilated (MV) patients in the intensive care unit (ICU) is essential for improving patients' hospitalization experiences and outcomes. However, numerous hospitals have reduced the visiting time and frequency in ICUs due to the global spread of SARS-CoV-2 in recent years, aggravating mental problems and reducing the satisfaction of ICU patients and their families. Therefore, we propose an effective intervention strategy to enhance patient-family bonding and improve patient mental health and ICU experience by constructing a remote cross-platform virtual reality collaboration system (VRCS) for connecting family members at home with patients in the ICU. We aim to assess the effects of VRCS on the mental health of ICU patients.

DETAILED DESCRIPTION:
Introduction: The ICU is a specialized medical unit equipped with state-of-the-art monitoring equipment and life support machines to provide care for critically ill patients. Patients in the ICU receive extensive and dynamic monitoring to ensure the timely and effective treatment to reduce mortality rates. However, despite the benefits of ICU care, patients may experience severe mental distress and poor hospital experiences due to a variety of factors. In fact, studies have shown that a majority of ICU patients (over 60%) experience long-lasting psychological problems. Current studies have shown that involving families in the care process can help patients feel more secure and lead to greater satisfaction among patients and their families. But due to nosocomial infection, most ICUs still adopt a restrictive visiting strategy. Therefore, we propose a virtual visiting method based on a remote cross-platform VR collaboration system (VRCS) to help patients get rid of the stressful ICU environments, and provide real-time interaction and communication between patients and their families, so as to improve the mental health and hospitalization experience of patients, as well as improve the satisfaction of patients and families.

Methods and Materials: This single-blind, randomized, controlled trial will be conducted from January to December 2023 in the ICU of Peking Union Medical College Hospital (PUMCH). We aim to randomize 566 adult ICU patients with an expected mechanical ventilation time over 24 hours into the VRCS intervention group and the control group (283 in each group). The patients in the VRCS group can see their families in a virtual natural forest environment through VR headsets and communicate with them through an eye-tracking interaction method. Simultaneously, their family members can see and communicate with the patients through smartphones, computers, or TVs at home. The primary objective is to study the effect of VRCS on the mental health and hospitalization experience of MV patients during the ICU stay. The secondary outcome is to assess the effect of VRCS on the incidence of delirium and the quality of patient-family communication during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation time > 24h, and is currently undergoing mechanical ventilation;
* Age ≥ 18 years old, no upper age limit;
* Language: Chinese;
* RAAS score ≥ -2 points;
* Hemodynamic stability.

Exclusion Criteria:

* Severe visual impairment (WHO classification: severe visual impairment) or hearing impairment (WHO classification: severe hearing loss);
* Cognitive and consciousness impairment;
* Head trauma or surgery resulting in an inability to wear HMDs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-03-17 (Estimated); Study Completion 2024-03-17 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | 1 year
  The HADS is designed by Zigmond and Snaith in 1983 to assess anxiety and depression symptoms in medical patients, including 14 items and every item scoring from 1 to 4. It includes two scales, one for anxiety (HADS-A) and another for depression (HADS-D). Each scale has 7 items and has a total score range from 7 to 28. The diagnostic criteria are that if the diagnosed person scores more than 11 points on any scale, it can be regarded as a confirmed case.

SECONDARY OUTCOMES:
Blood pressure | 1 year
  The blood pressure(mmHg) will be collected from a bedside monitor every 6 hours until 48 hours after the intervention. Both Systolic and Diastolic Blood Pressure will be measured.
Heart Rate | 1 year
  The heart rate(bpm) will be collected from a bedside monitor every 6 hours until 48 hours after the intervention.
Respiratory rate | 1 year
  The respiratory rate (breaths/min) will be collected from a bedside monitor every 6 hours until 48 hours after the intervention.
Oxygen saturation level | 1 year
  The oxygen saturation level (SpO2, %) will be collected from a bedside monitor every 6 hours until 48 hours after the intervention.
Activation of cranial nerve signals | 1 year
  The activation of cranial nerve signals will be collected from a bedside monitor every 6 hours until 48 hours after the intervention.
Number of Acute Cardiac Events | 1 year
  The number of acute cardiac events is assessed by analgesic drug dosage, which is recorded by the physicians and nurses.
Duration of Mechanical Ventilation | 1 year
  The duration of mechanical ventilation is daily recorded by the physicians and nurses.
ICU Days | 1 year
  The ICU stays are daily recorded by the physicians and nurses in ICU.
Patient Health Questionnaire-9 (PHQ-9) | 1 year
  It includes 9 items and every item is scored from 0 points to 3 points. Thus, the total score is range from 0 to 27 points. The higher the score, the more severe symptoms of the depression. Since the questionnaire relies on patient self-report, all responses should be verified by the clinician, and a definitive diagnosis is made on clinical grounds taking into account how well the patient understood the questionnaire, as well as other relevant information from the patient.
Positive and Negative Affect Schedule (PANAS) | 1 year
  It includes 20 items and each item is scored from 1 point to 5 points. The higher the score, the stronger the emotion. To score the positive effect, one would add up the scores on lines 1, 3, 5, 9, 10, 12, 14, 16, 17 & 19. Scores may range anywhere from 10 - 50. Higher scores represent higher levels of positive affect. Mean scores: momentary=29.7 and weekly=33.3. To score the negative emotions, one would add up the scores on items 2, 4, 6, 7, 8, 11, 13, 15, 18 & 20. Scores may range anywhere from 10 - 50. Higher scores represent higher levels of negative affect. Mean scores: momentary = 14.8 and weekly = 17.4.
Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) | 1 year
  The CAM-ICU is designed to monitor and evaluate the incidence of Delirium, which has four items ((1) altered mental status/fluctuating course, (2) inattention, (3) altered level of consciousness, and (4) disorganized thinking) and each item has two factors (positive or negative). The physicians can diagnose patients with delirium when the results of item (1), item (2), and item (3) / item (4) are positive. The CAM-ICU will be used after the while intervene.
Family In-Patient Communication Survey (FICS) | 1 year
  The FICS is designed by AM Torke et al. to measure the communication experiences of family members of hospitalized patients. It is comprised of 30 items (1-5 points) in which the individual rates how much they agree or disagree with each statement, while some items (indicated with an asterisk) are reverse scored. The first 18 items assess communication - information, while the final 12 items assess emotional support.
Family Satisfaction with Care in the Intensive Care Unit (FS-ICU) | 1 year
  The FS-ICU is designed by Heyland et al to evaluate the family satisfaction level. It can evaluate the family's satisfaction with care (FS-Care) and satisfaction with decision-making (FS-DM). The results include the calculated score on the total instrument (FS-Total) and the calculated scores for the 2 subscales (FS-Care & FS-DM).

CONTACTS AND LOCATIONS:
Overall Officials: Yun Long, MD, Study Director — Peking Union Medical College
Locations (1):
- PUMC, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No